CLINICAL TRIAL: NCT03028948
Title: Internet Intervention for Sun Protection and Skin Self-check Behaviors
Brief Title: Interactive Tailored Website to Promote Sun Protection and Skin Self-Check Behaviors in Patients With Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Virginia (Other)
Responsible Party: Principal Investigator, Sharon Manne, PhD, Professor and Associate Director of Population Science, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 131403; NCI-2017-00084 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2014000095 (Other: Rutgers, The State University of New Jersey); Pro2014000095 (Other: Rutgers Cancer Institute of New Jersey); R01CA171666 (NIH)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Stage 0 Skin Melanoma; Stage I Skin Melanoma; Stage IA Skin Melanoma; Stage IB Skin Melanoma; Stage II Skin Melanoma; Stage IIA Skin Melanoma; Stage IIB Skin Melanoma; Stage IIC Skin Melanoma; Stage III Skin Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (ITW) (Experimental): Patients access ITW and complete each module over 30-40 minutes. All patients in Phase II complete surveys over 20-40 minutes at 8, 24, and 48 weeks.
  Interventions: Other: Internet-Based Intervention; Other: Questionnaire Administration; Other: Survey Administration
- Arm II (usual care) (Active Comparator): Patients receive usual care and are then offered ITW. All patients in Phase II complete surveys over 20-40 minutes at 8, 24, and 48 weeks.
  Interventions: Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Access ITW
  Arms: Arm I (ITW)
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well an interactive tailored website works in promoting sun protection and skin self-check behaviors in patients with stage 0-III melanoma. An internet-based program may help individuals to perform skin self-checks and engage in sun protection behaviors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the impact of the interactive tailored website (ITW) versus usual care on skin self-examination (SSE) and sun protection behaviors among individuals diagnosed with melanoma.

SECONDARY OBJECTIVES:

I. To examine mediators of the impact of the intervention. The effects of the intervention on SSE and sun protection behaviors will be mediated by melanoma knowledge, self-efficacy for SSE and sun protection behaviors, perceived benefits of SSE and sun protection behaviors, perceived barriers to SSE and sun protection behaviors, and perceived controllability of melanoma.

TERTIARY OBJECTIVES:

I. To examine moderators of the impact of the intervention. To evaluate whether ITW effects are moderated by the following factors: time since diagnosis, disease stage, age, sex, income, education, Internet experience, distress about melanoma, worry about recurrence, and evaluation and usage of the ITW.

OUTLINE:

Phase I: Patients review draft website content materials in a semi-structured format and provide feedback via open- and closed-ended questions for the development, testing, and finalization of ITW.

Phase II: Patients are randomized into 1 of 2 arms.

ARM I: Patients access ITW and complete each module over 30-40 minutes.

ARM II: Patients receive usual care and are then offered ITW.

All patients in Phase II complete surveys over 20-40 minutes at 8, 24, and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Diagnosis of primary pathologic stage 0-III cutaneous malignant melanoma
* Phase I: From 3-36 months post-surgical treatment
* Phase I: Access to the internet
* Phase I: Able to speak and read English
* Phase I: Able to provide informed consent
* Phase II: Diagnosis of primary pathologic stage 0-III cutaneous malignant melanoma
* Phase II: From 3-24 months post-surgical treatment
* Phase II: Not adherent to thorough SSE (i.e., did not check every area of the body at least once during the past 2 months)
* Phase II: Not adherent to sun protection recommendations (i.e., mean score < 4 [which corresponds to "often"] on a 5-point scale [from 1 = "never" to 5 = "always"] that assesses the frequency of engaging in four sun protection behaviors)
* Phase II: Access to a computer connected to the internet
* Phase II: Able to speak and read English
* Phase II: Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Coups, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Coups EJ, Manne SL, Ohman Strickland P, Hilgart M, Goydos JS, Heckman CJ, Chamorro P, Rao BK, Davis M, Smith FO, Thorndike FP, Ritterband LM. Randomized controlled trial of the mySmartSkin web-based intervention to promote skin self-examination and sun protection behaviors among individuals diagnosed with melanoma: study design and baseline characteristics. Contemp Clin Trials. 2019 Aug;83:117-127. doi: 10.1016/j.cct.2019.06.014. Epub 2019 Jun 27. PMID 31255801

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 485 consented participants, 441 completed baseline survey and were randomized to treatment.
Groups:
- mySmartSkin: Of 485 enrolled individuals, 224 were randomized to MSS.
  These individuals access MSS content and complete the three educational Cores. Individuals completed surveys at baseline, 8 weeks, 24 weeks and 48 weeks.
- Usual Care: Of the 485 enrolled individuals, 217 were randomized to the UC condition.
  These participants received the usual clinical follow-up care. Individuals completed surveys at baseline, 8 weeks, 24 weeks and 48 weeks.
Period: 8 Week Follow-up
Arm/Group | mySmartSkin | Usual Care
Started | 224 | 217
Completed | 198 | 215
Not Completed | 26 | 2
Period: 24 Week Follow-up
Arm/Group | mySmartSkin | Usual Care
Started | 224 | 217
Completed | 189 | 207
Not Completed | 35 | 10
Period: 48 Week Follow-up
Arm/Group | mySmartSkin | Usual Care
Started | 224 | 217
Completed | 180 | 202
Not Completed | 44 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mySmartSkin | Usual Care | Total
Number analyzed (Participants) | 224 | 217 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (12.9) | 60.8 (13.7) | 61.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 113 | 216
  Male | 121 | 104 | 225
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 218 | 214 | 432
  Non-Hispanic Black | 1 | 0 | 1
  Non-Hispanic Other | 2 | 0 | 2
  Hispanic | 3 | 3 | 6
Level of Education [Count of Participants; unit: Participants]
  ≤ High school graduate | 32 | 22 | 54
  Some college | 42 | 45 | 87
  College graduate | 70 | 63 | 133
  Graduate degree | 80 | 87 | 167
Annual Household Income [Count of Participants; unit: Participants]
  ≤ $59,999 | 37 | 26 | 63
  $60,000 to $99,999 | 56 | 53 | 109
  $100,000 to $149,999 | 45 | 39 | 84
  ≥ $150,000 | 68 | 68 | 136
  Unknown | 18 | 31 | 49
Marital Status [Count of Participants; unit: Participants]
  Married/partnered | 179 | 172 | 351
  Not married/partnered | 45 | 45 | 90
Frequency of using the Internet [Count of Participants; unit: Participants]
  2 or fewer days/week | 13 | 13 | 26
  3 to 5 days/week | 13 | 12 | 25
  Once a day | 40 | 23 | 63
  2 to 3 times/day | 53 | 65 | 118
  4 or more times/day | 98 | 101 | 199
  Unknown | 7 | 3 | 10
Level of comfort using the Internet [Count of Participants; unit: Participants]
  Very uncomfortable | 10 | 9 | 19
  Somewhat uncomfortable | 15 | 8 | 23
  Neither comfortable nor uncomfortable | 16 | 11 | 27
  Somewhat comfortable | 50 | 49 | 99
  Very comfortable | 126 | 137 | 263
  Unknown | 7 | 3 | 10
Number of melanoma risk factors (range 0-8) [Mean (Standard Deviation); unit: risk factors] | 4.3 (1.7) | 4.4 (1.6) | 4.4 (1.6)
Time since melanoma surgery [Count of Participants; unit: Participants]
  3 to < 14 months | 108 | 116 | 224
  14 to 24 months | 116 | 101 | 217
Disease stage [Count of Participants; unit: Participants] — Disease stage refers to primary pathologic stage of cutaneous malignant melanoma that the participant was diagnosed with. In this study, stage 0 and I are considered early stage melanoma. Earlier stages are associated with better outcomes and less serious disease.
  Participants
    0 | 67 | 69 | 136
    I | 126 | 119 | 245
    II | 18 | 16 | 34
    III | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Sun Protection Behavior Index
Description: Participants rated how often they engaged in four behaviors when outside on a sunny day: wearing sun screen with an Sun Protection Factor ≥ 30, wearing a long-sleeved shirt, wearing a wide-brimmed hat, and staying in the shade. Items were rated on a five-point Likert scale (1=never, 2= rarely, 3= sometimes, 4= often, 5=always). In this case, higher values are associated with more protection behaviors. Subscales were averaged to compute the total index score.
Time Frame: At 24 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- mySmartSkin; Usual Care: Participants rated how often they engaged in four behaviors when outside on a sunny day: wearing sun screen with an Sun Protection Factor ≥ 30, wearing a long-sleeved shirt, wearing a wide-brimmed hat, and staying in the shade. Items were rated on a five-point Likert scale (1=never, 5=always).
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 189 | 207
scores on a scale | 3.54 (0.74) | 3.37 (0.84)

2. Primary Outcome: Number of Participants That Performed a Thorough Skin Self-examination (SSE) in the Past 2 Months
Description: Defined as thoroughly examining each area of the body during the most recent skin self-check in the last 2 months.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- mySmartSkin; Usual Care: Performance of a thorough SSE was defined as examining every area of the body during the most recent SSE. Participants reported if they had checked each part of their body for signs of cancer through a yes/no question response in the last 2 months and 6 months.
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 198 | 215
Participants
  Yes | 59 | 16
  No | 139 | 199

3. Secondary Outcome: Performance of Thorough Skin-self-examination (SSE) in the Past 4 Months
Description: Defined as thoroughly examining each area of the body during the most recent skin self-check in the past 4 months
Time Frame: At 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- mySmartSkin; Usual Care: Performance of a thorough SSE was defined as examining every area of the body during the most recent SSE. Participants reported if they had checked each part of their body for signs of cancer through a yes/no question response in the last 4 months.
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 189 | 207
Participants
  Yes | 54 | 24
  No | 132 | 182
  Unknown | 3 | 1

4. Secondary Outcome: Performance of Thorough Skin-self-examination (SSE) in the Past 6 Months
Description: Defined as thoroughly examining each area of the body during the most recent skin self-check in the past 6 months
Time Frame: 48 weeks
Measure: Count of Participants; unit: Participants
Groups:
- mySmartSkin; Usual Care: Performance of a thorough SSE was defined as examining every area of the body during the most recent SSE. Participants reported if they had checked each part of their body for signs of cancer through a yes/no question response in the last 6 months.
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 180 | 202
Participants
  Yes | 54 | 26
  No | 121 | 169
  Unknown | 5 | 7

5. Secondary Outcome: Number of SSEs Performed
Description: Total number of SSEs performed (regardless of their thoroughness)
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Number of Body Areas Examined
Description: Total number of body areas examined during the most recent SSE in the last 2 months
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Use of Tools to Facilitate SSE
Description: Use of a mirror, having someone else help, or using a body mole map during the most recent SSE
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Frequency of Engaging in Each Individual Sun Protection Behavior From the Sun Protection Behavior Index
Description: Frequency (from 1 = never to 5 = always) of wearing sunscreen with an SPF ≥ 30, wearing a long-sleeved shirt, wearing a wide-brimmed hat, and staying in the shade
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Number of Sunburns
Description: Total number of sunburns received
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Wearing Long Pants
Description: Frequency (from 1 = never to 5 = always) of wearing long pants
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Wearing Sunglasses
Description: Frequency (from 1 = never to 5 = always) of wearing sunglasses
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Sunbathing
Description: Frequency (from 1 = never to 5 = always) of spending time in the sun in order to get a tan
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Distress About Melanoma
Description: Level of distress (from 1 = not at all distressed to 10 = extremely distressed)
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Worry About Melanoma Recurrence
Description: Mean rating of four questions regarding worry about melanoma recurrence
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Perceived Risk of Melanoma Recurrence
Description: Mean rating of four questions regarding perceived risk of melanoma recurrence
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Biopsies Conducted
Description: Number of biopsies conducted
Time Frame: At 48 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Indoor Tanning
Description: Number of times indoor tanned in the past year
Time Frame: At 48 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Diagnosis of New or Recurrent Skin Cancers
Description: Whether a new or recurrent skin cancer was diagnosed
Time Frame: At 48 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Indicators of Study Feasibility
Description: Ineligibility rate and reasons, recruitment rate and reasons for refusal, differences in sociodemographic factors between study decliners and those recruited, dropout rate and reasons.
Time Frame: At 48 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Visits to Healthcare Provider Related to Skin Surveillance
Description: Receipt of a physician skin examination and the reason for the visit
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Impact and Effectiveness of the Interactive Tailored Website
Description: Perceived Internet Impact and Effectiveness Questionnaire was used. This 20-item survey was used to measure the degree to which MSS helped the participant learn how to be prepared to conduct SSE and engage in sun protection behaviors as well as feel in control of his/her health and feel less worried about melanoma. A Likert scale was used for each question (1=not at all, 2=slightly, 3=somewhat, 4=mostly, 5=very). The scores from each question were averaged to compute the total scale score for each participant. The total scores for each participant were also averaged to find the overall average across MSS participants. Higher values represent greater effectiveness of the program.
Time Frame: At 8 weeks
Population: This survey was only conducted among those who were randomized to MSS
Measure: Mean (Standard Deviation); unit: scores on scale
Groups:
- mySmartSkin: At the 8 week follow-up, participants enrolled in the MSS intervention completed a 20-item Impact and Effectiveness measure assessing the degree to which MSS helped the participant learn how to be prepared to conduct SSE and engage in sun protection behaviors as well as feel in control of his/her health and feel less worried about melanoma (1=not at all, 5=very).
- Usual Care: Did not complete.
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 198 | 0
scores on scale | 4.1 (0.72) |

22. Other Pre Specified Outcome: Usage of the Interactive Tailored Website
Description: Number of visits to the website, the number of monthly skin self-checks completed, the number of updates to the sun-safe action plan, and starting/completing the remaining sections of the website (Introduction; Getting Ready to Do a Skin Self-Check; Practice Sun-Safe Behaviors).
Time Frame: At 8, 24 and 48 weeks
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Evaluation and Utility of the Interactive Tailored Website
Description: Internet Evaluation and Perceived Utility Questionnaire and the Internet Adherence Questionnaire was used. This 15-item survey assessed the program characteristics, including usefulness, convenience, ease of use, worry about privacy, ease of navigation, and satisfaction with the program. A Likert scale was used for each question (1=not at all, 2=slightly, 3=somewhat, 4=mostly, 5=very). The scores from each question were averaged to compute the total scale score for each participant. The total scores for each participant were also averaged to find the overall average across MSS participants. Higher values represent higher scores in terms of utility and evaluation of the program.
Time Frame: At 8 weeks
Population: Only the participants randomized to the intervention arm completed this survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- mySmartSkin: At the 8 week follow-up, participants enrolled in the MSS intervention completed a 15-item Evaluation and Utility survey, which assessed program characteristics, including usefulness, convenience, ease of use, worry about privacy, ease of navigation, and satisfaction with the program (1=not at all, 5=very).
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 198 | 0
scores on a scale | 4.3 (0.65) |

24. Secondary Outcome: Sun Protection Behavior Index
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 224 | 217
scores on a scale | 3.25 (.75) | 3.29 (.76)

25. Secondary Outcome: Sun Protection Behavior Index
Description: as for outcome 1
Time Frame: At 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 198 | 215
scores on a scale | 3.4 (.78) | 3.31 (.81)

26. Secondary Outcome: Sun Protection Behavior Index
Description: as for outcome 1
Time Frame: At 48 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | mySmartSkin | Usual Care
Number analyzed (Participants) | 179 | 202
scores on a scale | 3.65 (.72) | 3.52 (.79)

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored/assessed
Description: Adverse events were not monitored/assessed. There is no risk for participating in this study and, therefore, zero participants are at risk of facing an adverse event.
Arm/Group | mySmartSkin | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Findings may be less generalizable to those with low sun protection behavior. We recruited from one state so participant pool may not represent the US population. SSE and sun protection were assessed using self-report. Sun content was in the last core and reviewed by fewer participants. Sample was primarily non-Hispanic white.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT03028948/Prot_SAP_001.pdf
  • Informed Consent Form (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03028948/ICF_000.pdf